CLINICAL TRIAL: NCT01770470
Title: A Pilot Study of Dietary Chitosan Chewing Gum in Dialysis Patients
Brief Title: Chitosan Chewing Gum Study in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Other Study IDs: HP-00045129
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: End Stage Renal Disease
Keywords: serum phosphate; chitosan; kidney disease; salivary phosphate
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases | interventions — Chitosan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving chronic hemodialysis: Dialysis patients chewing chitosan-containing gum
  Interventions: Dietary Supplement: Chitosan

INTERVENTIONS:
Dietary Supplement: Chitosan — The product chitosan is contained in a chewing gum formulation

SUMMARY:
The purpose of the pilot study is to determine the impact of short-term administration of chitosan-containing chewing gum on phosphate levels in patients with elevated serum phosphate levels.

DETAILED DESCRIPTION:
The impact of using salivary phosphate binders in ESRD patients is not fully known. The purpose of the pilot study is to determine the impact of short-term administration of chitosan-containing chewing gum on phosphate levels in patients with elevated serum phosphate levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years old
* ESRD receiving hemodialysis
* serum phosphate > 6.0 mg/dL

Exclusion Criteria:

* Unable to sign consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Outpatient hemodialysis facility
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Serum phosphate | 6 weeks
  Serum phosphate will be drawn 3 times per week over 2 weeks (during gum therapy), then once at 4 weeks and once at 6 weeks.

SECONDARY OUTCOMES:
Salivary phosphate levels | 6 weeks
  Salivary phosphate will be assessed 3 times per week over 2 weeks (during gum therapy), then once at 4 weeks and once at 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dowling, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States